CLINICAL TRIAL: NCT00166829
Title: The Effect of Sirolimus on the Pharmacokinetics of Tacrolimus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 920606
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2007-03-08 (Estimated); Status verified 2003-08

CONDITIONS: Kidney Transplantation
Keywords: Tacrolimus; Sirolimus; Mycophenolic acid; Immunosuppressive Agents; Immunosuppression; Kidney Transplantation; Transplantation
MeSH Terms: interventions — Sirolimus; Tacrolimus; Mycophenolic Acid

INTERVENTIONS:
Drug: sirolimus, tacrolimus, mycophenolate mofetil

SUMMARY:
The purpose of this study is to understand whether the pharmacokinetics of tacrolimus is influenced by the concurrent use of sirolimus.

DETAILED DESCRIPTION:
The controlled clinical trial held in NTUH in 2001 revealed that the bioavailability of tacrolimus when combined with sirolimus is lower than that reported in the literature where tacrolimus was not combined with sirolimus. To determine if the difference was due to the drug interaction between sirolimus and tacrolimus, a controlled clinical trial was proposed.

The purpose of this study is to understand whether the pharmacokinetics of tacrolimus is influenced by the concurrent use of sirolimus.

ELIGIBILITY:
Inclusion Criteria:

* De novo kidney transplant patients
* Aged 13 - 65 years
* Having aminotransferase concentrations within 2 times the upper limit of normal

Exclusion Criteria:

* Pregnancy
* Tuberculosis
* Hepatitis B or C carrier status
* Human immunodeficiency virus-positive status
* Retransplantation or multi-organ transplantation
* History of rheumatoid arthritis

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2004-05

PRIMARY OUTCOMES:
The influence of sirolimus on the pharmacokinetics of tacrolimus in renal transplant patients

SECONDARY OUTCOMES:
Compare the outcome of tacrolimus/sirolimus and tacrolimus/mycophenolate in rejection prevention

CONTACTS AND LOCATIONS:
Overall Officials: Po-Huang Lee, MD, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Tsai MK, Wu FL, Lai IR, Lee CY, Hu RH, Lee PH. Decreased acute rejection and improved renal allograft survival using sirolimus and low-dose calcineurin inhibitors without induction therapy. Int J Artif Organs. 2009 Jun;32(6):371-80. doi: 10.1177/039139880903200608. PMID 19670189